CLINICAL TRIAL: NCT06966960
Title: Online RPG Interactive Adventure Games Combined With an E-book Learning Mode to Enhance Nursing Students' Motivation and Effectiveness in Learning Obstetric Fetal Heart Rate Monitoring Technology
Brief Title: Online RPG Interactive Adventure Games Combined With an E-book Learning Obstetric Fetal Heart Rate Monitoring Technology
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ting-Shan Chang, Assistant Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CMUH114-REC2-028
Record Dates: First submitted 2025-04-26; First posted 2025-05-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Nursing Education Research
Keywords: fetal heart rate; e-book; nursing education; role-playing game; learning motivation; nursing

STUDY DESIGN:
Intervention Model Description: The study design will adopt a randomized controlled trial with repeated measures. A 60-minute intervention has been developed.
  Block randomization stratified by gender will be used, and eligible participants will be randomly assigned to either the experimental or control group in a 1:1 ratio using Random Allocation Software.
  Research assistants will code group assignments ("Group 1" and "Group 2") according to the randomization list, place the assignments into opaque sealed envelopes, and arrange them sequentially.
  On the day of the study, envelopes will be distributed in the order participants submit their consent forms. Participants will open the envelope themselves to learn their group assignment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online RPG interactive adventure game and e-book (Experimental): Integration of online RPG interactive adventure games with an e-book learning mode for the instruction of obstetric fetal heart rate monitoring technology.
  Interventions: Behavioral: Online RPG adventure games and e-book learning.
- e-book (Active Comparator): E-book learning mode for obstetric fetal heart rate monitoring technology.
  Interventions: Behavioral: E-book

INTERVENTIONS:
Behavioral: Online RPG adventure games and e-book learning. — Learning obstetric fetal heart rate monitoring technology through online RPG adventure games and e-book learning.
  Arms: Online RPG interactive adventure game and e-book
Behavioral: E-book — E-book learning mode for obstetric fetal heart rate monitoring technology.
  Arms: e-book

SUMMARY:
One of the main goals of nursing education is to cultivate essential clinical skills in students to ensure they can provide safe, effective, and compassionate care within a medical environment. In the field of obstetric nursing, the precise mastery of fetal heart rate monitoring is crucial as it significantly impacts the students' future ability to assess the health conditions of both the mother and the fetus in clinical settings. This becomes increasingly important in today's context of declining birth rates. However, traditional nursing education, which mainly relies on knowledge transmission and simulation demonstrations, not only struggles to stimulate students' interest but often leads to ineffective learning outcomes. With the rapid advancement of technology, these limitations no longer meet the current needs of nursing education and students. Therefore, this study proposes to build and explore a new teaching model based on the ARCS motivation theory, integrating online role-playing games (RPGs) and interactive e-books to enhance nursing students' learning motivation and effectiveness.

DETAILED DESCRIPTION:
This research project is planned over two years. The first year will focus on developing entertaining, interactive, and context-rich RPGs and e-books to enhance learning relevance and attention. By designing a tiered challenge system, not only will successful experiences be created, but students' confidence will also be bolstered. Additionally, an effective feedback mechanism will be set up to enhance the satisfaction of learning. The second year will involve a randomized controlled trial to validate the learning outcomes and motivation of nursing students in mastering fetal heart rate monitoring techniques. the design of the RPGs and e-books will be optimized to enhance the learning effectiveness and motivation of newly qualified nurses in real clinical settings, and extended to clinical education, aiming to fill the gaps in current educational models and improve the quality of nursing care.

This project establishes new digital materials and learning models for a commonly used skill in obstetric care. The research outcomes will help develop flexible, personalized learning pathways, enabling students to learn autonomously anytime, anywhere. This innovative approach not only enhances students' learning motivation and adds a new dimension to both teaching and self-study materials but also aids in their better application in clinical practice, thereby increasing the safety and efficiency of clinical care. Moreover, the application of this model offers a fresh perspective and approach to nursing education, promoting its ongoing development and quality enhancement.

ELIGIBILITY:
Inclusion Criteria:

1. It is expected to include 100 people.
2. Age 20 to 30 years old.
3. A third-year nursing student.
4. Completed basic nursing studies.
5. Agree to participate in this study and sign the research consent form.

Exclusion Criteria:

1. Students who were scheduled to take a leave of absence at the time of data collection.
2. No basic nursing training has been taken.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2025-10-14 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
Fetal Heart Rate Monitoring and Nursing Knowledge Questionnaire | The experimental group and the control group will Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  The questionnaire consists of 10 items. Each correct answer is awarded 10 points, and each incorrect answer is awarded 0 points. The total score ranges from 0 to 100 points. The items, preliminarily developed, include clinical scenario-based questions in a multiple-choice format, primarily focusing on the interpretation of fetal heart rate monitoring and corresponding nursing interventions based on the interpretation results.
Fetal Heart Rate Monitoring and Nursing Skills Assessment Scale | The experimental group and the control group will Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  This outcome is assessed using the "Fetal Heart Rate Monitoring and Nursing Skills Assessment Scale," which includes 12 items covering domains such as professional attitude, patient identification, explanation of monitoring purpose, hand hygiene, and the correct step-by-step application of fetal monitoring equipment. The total score ranges from 0 to 100, with higher scores indicating better skill performance.
  Time Frame: Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  Unit of Measure:
  Score on a 0-100 scale
Fetal Heart Rate Monitoring and Nursing Self-Efficacy Scale | The experimental group and the control group will Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  This outcome is assessed using the "Fetal Heart Rate Monitoring and Nursing Self-Efficacy Scale," consisting of 10 items rated on a 4-point Likert scale. Participants evaluate their own ability to perform related tasks, where 1 = insufficient ability and 4 = expert ability. The total score ranges from 10 to 40, with higher scores indicating greater self-efficacy in performing fetal heart monitoring and related nursing skills.
  Time Frame:
  Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  Unit of Measure:
  Total score on a 10-40 scale
ARCS-Based Learning Motivation Scale | The experimental group and the control group will Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  The scale assesses learners' motivation toward the educational materials across four dimensions: Attention (12 items), Relevance (9 items), Confidence (9 items), and Satisfaction (6 items), for a total of 36 items. Responses are rated on a 5-point Likert scale, ranging from 5 ("Strongly Agree") to 1 ("Strongly Disagree"). The total score ranges from 36 to 180 points, with higher scores indicating stronger learning motivation.
Critical Thinking Disposition Scale | The experimental group and the control group will Baseline (prior to intervention), immediately after intervention, and 4 weeks after intervention
  This scale consists of 20 items and adopts a 6-point Likert scoring method: 1 (Never), 2 (Almost Never), 3 (Rarely), 4 (Sometimes), 5 (Often), and 6 (Always). It measures critical thinking disposition, which refers to an individual's tendency to engage in systematic analysis, maintain an open-minded attitude with empathy, and possess a wise curiosity for questioning, integration, and reflection, all of which facilitate critical thinking processes.

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Shan Chang, Assistant Professor, Principal Investigator — China Medical University, Taiwan
Locations (1):
- China Medical University, Taichung, Taiwan, Taiwan